CLINICAL TRIAL: NCT05266521
Title: Safety and Efficacy Assessment of Using the zLOCK Facet Stabilization System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZygoFix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMS
Record Dates: First submitted 2022-02-13; First posted 2022-03-04 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain
Keywords: Stabilization; Facet arthritis; Spondylolisthesis; Stenosis
MeSH Terms: conditions — Low Back Pain; Spondylolisthesis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zLock Facet Locking Implant System (Experimental): Device: zLOCK Facet Stabilization System zLOCK Facet Stabilization System is a device intended to provide posterior stability in lumbar spine in order to reduce lumbar back pains
  Interventions: Device: zLOCK Facet Stabilization System

INTERVENTIONS:
Device: zLOCK Facet Stabilization System — zLOCK Facet Stabilization System is a device intended to provide posterior stability in lumbar spine in order to reduce lumbar back pains

SUMMARY:
The zLOCK Facet Stabilization System is a fixation device intended to provide posterior stability in the lumbar spine fusion procedure. The system can be placed either as an adjunct to an inter-vertebral anterior cage or as stand-alone with/ without additional decompression of the dural sac or nerve roots as appropriate for the specific patient and surgeon's discretion. The zLOCK implant is placed inside the facet to stabilize the motion and enhance the bony fusion of the joint. The zLOCK Facet Stabilization System is intended for single-level stabilization of a spinal motion segment in order to promote bony fusion of the joint. The zLOCK system is indicated for use from L1-L2 to L5-S1 joints.

The zLOCK implant is inserted into the facet joint space while adapting to the joint's changing geometry. Stabilization is achieved by a firm grip of each joint bone and resisting any relative motion. The zLOCK implant is placed percutaneously and requires only one incision per side, thereby reducing the invasiveness procedure duration and shortening the recovery period.

This pivotal study was designed in order to assess the safety and effectiveness of the zLOCK system.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is scheduled for spine surgery with at least one of the following:

   * Degenerative Spondylolisthesis grade 1;
   * Mild to Moderate stenosis;
   * Degeneration of the facets.
2. When used stand-alone disc height should be maximum 50% of the adjacent disc height.
3. 18< Age <75
4. Weight < 100Kg
5. Signed informed consent form
6. At least 3 months of unsuccessful conventional treatments

Exclusion Criteria:

1. Fusion procedure performed or required in more than one motion segment.
2. Acute or chronic spinal infections.
3. Osteoporosis when used in adjunct to an anterior interbody cage (DEXA < -2.5).
4. Absence of posterior spinal elements including the pedicle, pars interarticularis, facet joints, spinous process and the majority of the lamina which make it unstable or not possible to place.
5. Any entity or conditions that totally preclude the possibility of fusion, i.e. cancer or kidney dialysis.
6. Obesity (BMI ≥30)
7. Unilateral application of device, except in combination with anterior interbody cages.
8. Known sensitivity to Titanium.
9. Alcoholism, or drug abuse
10. Subject with a cardiac pacemaker or other implanted electro medical device
11. Women who are either pregnant or nursing at the time of screening (to be verified by test in case of woman of child-bearing potential that do not practice medically acceptable methods of contraception)
12. Concurrent participation in another clinical trial using any investigational drug or device.
13. Mental disorders.
14. Tumor
15. Fracture or other instabilities of the posterior elements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-07 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by paucity of device related reoperation | 3 months
  The safety of the zLOCK Facet Implant System will be established based on the paucity of device-related reoperations.

SECONDARY OUTCOMES:
Change in pain level measured by Visual Analog Score for pain | 1 year
  The efficacy assessment of the ZygoFix Facet stabilization System will be established by change in pain level
  .

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Levy, Dr., Study Director — ZygoFix
Locations (2):
- MedizinischenFakultät der Universität Rostock, Rostock, Germany
- AOU Policlinico "Paolo Giaccone", Palermo, Italy

IPD SHARING:
Plan to Share IPD: No